CLINICAL TRIAL: NCT04795713
Title: A Phase 1 Open-label, Multicenter, Dose-ranging Study to Investigate Safety and Tolerability, Efficacy, Pharmacokinetics, Pharmacodynamics and Immunogenicity of MT-6402 in Subjects With Advanced Solid Cancer That Expresses PD-L1
Brief Title: Study of MT-6402 in Subjects With Advanced Solid Cancer That Expresses PD-L1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated by Sponsor
Sponsor: Molecular Templates, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MT-6402-001
Record Dates: First submitted 2021-02-08; First posted 2021-03-12 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumor; Non-small Cell Lung Cancer; Squamous Cell Carcinoma of Head and Neck
Keywords: PD-L1 Positive; Relapsed or Refractory; Prior PD-1 or PD-L1 treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PD-L1 Positive NSCLC (Experimental): Subjects with PD-L1 Positive Lung Carcinoma (NSCLC) who received prior PD-1/PD-L1 treatment
  Interventions: Drug: MT-6402
- PD-L1 Positive SCCHN (Experimental): Subjects with PD-L1 Positive Squamous Cell Carcinoma of the head and neck (SCCHN), refractory to or ineligible for platinum-based therapy, who received prior PD-1/PD-L1 treatment
  Interventions: Drug: MT-6402
- Other relapsed/refractory PD-L1 positive solid tumors (Experimental): Subjects with any other relapsed or refractory PD-L1 positive solid tumor who received PD-1/PD-L1 treatment.
  Interventions: Drug: MT-6402
- PD-L1 positive advanced cancer (Experimental): Subjects with PD-L1 positive advanced cancer (solid tumors)
  Interventions: Drug: MT-6402

INTERVENTIONS:
Drug: MT-6402 — Experimental Treatment

SUMMARY:
This will be a Phase 1 Open-label, dose escalation and expansion study of MT-6402 (an Engineered Toxin Body (ETB)) in subjects with advanced solid cancer that expresses PD-L1

DETAILED DESCRIPTION:
This study will be conducted in two sequential parts:

* Part 1 (Dose Escalation): The purpose of Part 1 is to evaluate the safety and tolerability of MT-6402 in subjects with advanced cancer (solid tumors) and to estimate the maximum tolerated dose (MTD)
* Part 2 (Dose Expansion): The purpose of Part 2 is to confirm the recommended Phase 2 dose (RP2D) and to evaluate the efficacy of MT-6402 in subjects with advanced cancer. Part 2 will include subjects with PD-L1 positive non-small cell lung cancer (NSCLC) who received prior PD-1/PD-L1 treatment, subjects with PD-L1 positive squamous cell cancer of the head and neck (SCCHN) who are refractory to or ineligible for platinum-based therapy and received prior PD-1/PD-L1 treatment and subjects with any other relapsed or refractory PD-L1 positive solid tumor who received PD-1/PD-L1 treatment.

Up to 138 eligible subjects will be identified and treated through competitive enrollment at multiple study centers

In Parts 1 and 2, a subject may participate for the following four (4) periods:

* Screening Period - up to 28 days before first dose of MT-6402
* Treatment Period - active period where a subject will receive doses of MT-6402 over a 28-day treatment period
* Short-term Follow-up Period - up to 90 days after last dose of MT-6402
* Long-term follow-up Period - up to 24 months after last dose of MT-6402

MT-6402 will be given as an intravenous (IV) infusion over 30 minutes on the same day every week (i.e., days 1, 8, 15 and 22) of each cycle. A cycle is defined as 28 days. A subject can continue receiving MT-6402 as long as it is well-tolerated or until the subject decides they no longer want to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

Part A

1. Subject must be at least 18 years old and must have histologically confirmed, unresectable, locally advanced, or metastatic PD-L1-expressing solid cancer not amenable to standard treatment, or for whom standard treatment is not available, or in the Investigator's opinion the standard treatment would not be in the subject's best interest. Any level of PD-L1 expression assessed by using any Food and Drug Administration (FDA) approved PD-L1 immunohistochemistry (IHC) assay is accepted. In addition, another PD-L1 assay may be considered acceptable if approved by the Medical Monitor. The assessment should have been performed on the most recent available tissue from a site of metastatic disease (if possible).
2. Subject must have evaluable or measurable disease.

   Part B
3. Requirements for separate cohorts enrolled in Part B are as follows:

   * Cohort 1: Histologically confirmed recurrent or metastatic NSCLC not amenable to standard treatment, or standard treatment is not available, or in the Investigator's opinion the standard treatment would not be in the subject's best interest. NOTE: subjects with driver mutations are only eligible if they have received all appropriate targeted therapies.
   * Cohort 2: Histologically confirmed recurrent, resistant, or metastatic SCCHN (oral cavity, oropharynx, hypopharynx, or larynx) not amenable to standard treatment, or standard treatment is not available, or in the Investigator's opinion the standard treatment would not be in the subject's best interest. Subjects who refuse radical resection are eligible. NOTE: nasopharyngeal cancer, squamous cell carcinoma of any other primary anatomic location in the head and neck, subjects with SCCHN of unknown primary, and subjects with skin squamous cell carcinoma (SCC) of the head and neck are not eligible for this arm. The tumor must be platinum resistant or the subject ineligible for platinum therapy due to hypersensitivity or concerns with ototoxicity.
   * Cohort 3: Subjects with any other relapsed or refractory PD-L1 positive solid tumor not amenable to standard treatment, or standard treatment is not available, or in the Investigator's opinion the standard treatment would not be in the subject's best interest, who received PD-1/PD-L1 treatment. Subjects with PD-L1 positive solid tumor types, for which PD-1/PD-L1 treatment is not approved, could be enrolled at the Investigator's discretion and after discussion with the Medical Monitor.
4. Positive PD-L1 expression as assessed by an FDA approved PD-L1 IHC assay is required. The assessment should have been performed on the most recently available tissue and form a site of metastatic disease (if possible). Subjects without PD-L1 measured by an FDA-approved diagnostic must have PD-L1 expression confirmed by an FDA-approved diagnostic on either archived tissue or a fresh biopsy. Subjects for whom PD-L1 expression has not been determined and do not have archived tissue will require a fresh biopsy for PD-L1 determination by an FDA-approved diagnostic.
5. Subjects must be willing to have a total of 2 on trial biopsies: one at baseline and the other within the last 2 weeks of Cycle 2. Subjects who required a fresh biopsy at screening may utilize the screening biopsy tissue in lieu of the baseline biopsy.
6. Subject must have at least 1 measurable tumor lesion according to RECIST 1.1.

   Parts A and B
7. Subject must have Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1.
8. Prior treatment must include a CPI (i.e., PD-1 inhibitors, PD-L1 inhibitors with or without CTLA-4 inhibitors) if there is an approved CPI for the specific cancer type. Subjects may also have received CPIs in an investigational setting. Subjects who have not received a CPI and where there is no approved CPI for the specific cancer type could be enrolled at the Investigator's discretion and after discussion with the Medical Monitor.
9. Subject must have adequate bone marrow function (NOTE: administration of blood products and growth factors is not allowed within 2 weeks prior to screening laboratory tests):

   * absolute neutrophil count (ANC) ≥ 1,500/μL
   * platelet count ≥ 100,000/μL
   * hemoglobin ≥ 8.0 g/dL
10. Subject must have adequate renal function, based on estimated creatinine clearance (eCrCl) ≥ 50 mL/min, calculated by the Cockcroft-Gault equation.

    NOTE: At the Investigator's discretion, the eCrCl result < 50 mL/min may be verified by measured creatinine clearance (mCrCl) based on the 24-hour urine collection. Subjects with mCrCl ≥ 50 mL/min will be eligible irrespective of the eCrCl result calculated by the Cockcroft-Gault equation.
11. Subject must have adequate hepatic function, as determined by:

    * total bilirubin (or direct bilirubin for subjects with Gilbert's disease) < 1.5 × upper limit of normal (ULN)
    * aspartate aminotransferase (AST) ≤ 3 × ULN (or ≤ 5 × ULN if liver metastasis)
    * alanine aminotransferase (ALT) ≤ 3 × ULN (or ≤ 5 × ULN if liver metastasis)
12. Subject must have adequate serum albumin (albumin ≥ 2.5 g/dL)
13. Subjects capable of having children must have a negative highly sensitive pregnancy test within 72 hours before the start of treatment. Subjects who are postmenopausal (> 1 year since last menstrual cycle) or permanently sterilized (e.g., bilateral tubal occlusion, hysterectomy, bilateral salpingectomy) may be considered as not of reproductive potential.
14. Subjects of reproductive potential must agree either to abstain continuously from heterosexual intercourse or to use a highly effective birth control method from signing the informed consent until 30 days after the last dose of MT-6402 for subjects capable of bearing children and until 90 days after the last dose of MT-6402 for subjects capable of fathering children.

Exclusion Criteria:

Part A

1. Subjects without available tissue from a site of metastatic disease or easily biopsied lesion (biopsy sites of non significant risk, in the opinion of the Investigator) or unwilling to consent to biopsy.

   Part B
2. Subjects without easily biopsied lesions (biopsy sites of non significant risk, in the opinion of the Investigator) or unwilling to consent to baseline and end of Cycle 2 biopsy. Patients for whom a biopsy is not feasible must be discussed with the Medical Monitor.
3. Subjects unwilling to have baseline and on-study core biopsy (last 2 weeks of Cycle 2) performed.

   Parts A and B
4. History or current evidence of another neoplastic disease, except cervical carcinoma in situ, superficial noninvasive bladder tumors, curatively treated Stage I to II non melanoma skin cancer or any previous cancer curatively treated > 2 years before the start of treatment.
5. Active autoimmune disease currently under treatment or required systemic treatment within 2 years (replacement therapy, e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency is allowed). Subjects who have not required systemic treatment of an auto-immune disease for at least 2 years may be enrolled if permission is provided after discussion with the Medical Monitor.
6. Ongoing > Grade 1 immune related toxicity caused by prior CPI therapy (i.e., PD-1 inhibitors, PD-L1 inhibitors, or CTLA-4 inhibitors). Subjects with stable endocrinological AEs, e.g., hypothyroidism, adrenal insufficiency, hypopituitarism, or diabetes mellitus, must have been on a stable dose of supplemental therapy for at least 2 weeks before screening to be eligible for this study. History of repeat Grade 2 pneumonitis or carditis on previous CPI and/or Grade 3 immune related adverse event on previous CPI treatment.
7. Evidence of active noninfectious ≥ Grade 2 pneumonitis or current evidence of ≥ Grade 3 other underlying pulmonary disease.
8. Received any of the following PD-L1 inhibitors within the following time periods prior to the first dose of MT-6402: atezolizumab - 12 months; durvalumab - 7 months; avelumab - 2 months.
9. Any concurrent cancer treatment, apart from local treatment of non-target lesions for palliative intent (e.g., local surgery or radiotherapy).
10. Prior radiation therapy within 4 weeks before the start of study treatment. NOTE: A lesion in a previously irradiated area can only be considered target lesion if there has been radiographical disease progression since the end of radiation therapy.
11. Received approved or investigational treatment for the disease under study (except PD L1 inhibitors where exclusion criterion 6 applies) within 4 weeks before the start of treatment. For small molecules (MW < 0.9 kDa), the washout is 5 half-lives, but at least 2 weeks.
12. Subjects who have had allogeneic tissue or solid organ transplantation.
13. Current evidence of new or growing central nervous system (CNS) metastases during screening. Subjects with known asymptomatic CNS metastases will be eligible if they meet all the following criteria:

    1. Evidence of leptomeningeal metastasis.
    2. Have stable CNS disease on the computed tomography (CT) or magnetic resonance imaging (MRI) scan within 4 weeks before screening compared with prior neuro imaging.
14. Major surgical procedure (as defined by the Investigator) within 28 days prior to the start of study treatment.
15. History or current evidence of significant cardiovascular disease before the start of treatment, including but not limited to the following conditions:

    1. Angina pectoris requiring anti-anginal medication, (chest pain: Common Terminology Criteria for Adverse Events [CTCAE] Grade ≥ 2)
    2. Clinically significant valvular disease.
    3. Myocardial infarction within 12 months prior to the start of treatment.
    4. Arterial thrombosis or pulmonary embolism within 3 months before the start of treatment.
    5. History of Grade ≥ 2 symptomatic congestive heart failure (CHF) or New York Heart Association (NYHA) criteria Class ≥ II.
    6. Left ventricular ejection fraction (LVEF) < 55%, assessed preferably by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan if ECHO is not available, within 28 days before starting study treatment.
    7. High-risk uncontrolled arrhythmias (i.e., atrial tachycardia with a heart rate > 100/min at rest and upon repeated testing, significant ventricular arrhythmia (CTCAE Grade ≥ 2 [ventricular tachycardia], or higher-grade atrioventricular [AV]-block [second degree AV-block Type 2 [Mobitz 2] or third-degree AV-block]) or left ventricular bundle branch block. Subjects receiving digoxin, calcium channel blockers, or beta adrenergic blockers are eligible at the Investigator's discretion after consultation with the Medical Monitor if the dose has been stable for ≥ 2 weeks before the start of treatment with MT-6402.
    8. Any of the following within 3 months before the start of treatment: pericarditis (any CTCAE Grade), pericardial effusion (CTCAE Grade ≥ 2), non-malignant pleural effusion (CTCAE Grade ≥ 2) or malignant pleural effusion (CTCAE Grade ≥ 3) (subjects with pleural effusion that is manageable and stable > 3 months prior to study are eligible).
    9. QT interval correction for heart rate using Fridericia's formula (QTcF) ≥ 470 ms (average from 3 QTcF values on the triplicate 12-lead electrocardiogram [ECG]) at screening. In subjects with right bundle branch blocks, additional corrections will be performed to calculate the QT equivalent JT, and depending on the result the subject may be eligible with the agreement of the Medical Monitor.
16. Current evidence of uncontrolled human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) at screening. Serology testing is not required if seronegativity is documented in the medical history, and if there are no clinical signs suggestive of HIV or hepatitis infections, or suspected exposure. The following exceptions apply for subjects with positive viral serology:

    1. Subjects with HIV and an undetectable viral load and CD4 + T-cell (CD4+) counts ≥ 350 cells/mL may be enrolled, but must be taking appropriate opportunistic infection prophylaxis, if clinically relevant.
    2. Subjects with positive HBV serology are eligible if they have an undetectable viral load and the subject will receive antiviral prophylaxis for potential HBV reactivation per institutional guidelines.
    3. Subjects with positive HCV serology are eligible if quantitative polymerase chain reaction (PCR) for plasma HCV RNA is below the lower limit of detection. Concurrent antiviral HCV treatment per institutional guidelines is allowed.
17. Current treatment requiring systemic steroids at doses > 10 mg/day prednisone equivalent.
18. Subjects with a history of hypersensitivity or serious toxic reactions to kanamycin or other aminoglycosides.
19. Subjects with unintentional weight loss > 10% of their body weight over the preceding 2 months or less before screening.
20. Subjects who are pregnant or breastfeeding.
21. History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the Investigator or Medical Monitor, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of MT-6402 in subjects with advanced cancer (solid tumors) and to estimate the maximum tolerated dose (MTD) | 28 days (Part 1)
  Safety as measured by number of subjects with incidence of adverse events using CTCAE v4.0
Evaluate the tolerability of MT-6402 in subjects with advanced cancer (solid tumors) and to estimate the maximum tolerated dose (MTD) | 28 days (Part 1)
  Tolerability as measured by incidence of adverse events using CTCAE v5.0 and incidence of laboratory abnormalities
Confirm the recommended Phase 2 dose (RP2D) | 28 days (Part 2)
  Incidence of Adverse Events (AEs)
Evaluate efficacy of MT-6402 in subjects with advanced cancer by objective response rate (ORR) with RECIST 1.1 | up to 2 years (Part 2)
  ORR using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria

SECONDARY OUTCOMES:
Characterize the PK profile of MT-6402 in subjects with advanced cancer | up to 2 years (Parts 1 and 2)
  Maximum observed plasma concentration (Cmax)
Characterize the PK profile of MT-6402 in subjects with advanced cancer | up to 2 years (Parts 1 and 2)
  Time of maximum observed plasma concentration (tmax)
Characterize the PK profile of MT-6402 in subjects with advanced cancer | up to 2 years (Parts 1 and 2)
  Area under the concentration-time curve (AUC) from time zero to the last measurable concentration (AUC0-t)
Characterize the PK profile of MT-6402 in subjects with advanced cancer | up to 2 years (Parts 1 and 2)
  Interpolated AUC to infinity (AUC0-∞)
Characterize the PK profile of MT-6402 in subjects with advanced cancer | up to 2 years (Parts 1 and 2)
  Clearance (CL)
Characterize the PK profile of MT-6402 in subjects with advanced cancer | up to 2 years (Parts 1 and 2)
  Volume of distribution of steady-state (Vss)
Evaluate efficacy of MT-6402 in subjects with advanced cancer by ORR with RECIST 1.1 | up to 2 years (Part 1)
  ORR using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
Assess additional efficacy parameters | up to 2 years (Parts 1 and 2)
  Duration of response (DOR)
Assess additional efficacy parameters | up to 2 years (Parts 1 and 2)
  Progression-free survival (PFS)
Assess additional efficacy parameters | up to 2 years (Parts 1 and 2)
  Disease Control Rate (DCR)
Evaluate the immunogenicity of MT-6402 in subjects with advanced cancer | 28 days (Parts 1 and 2)
  Anti-drug antibodies (ADA)

OTHER OUTCOMES:
Evaluate the immunogenicity of MT-6402 in subjects with advanced cancer | 28 days (Parts 1 and 2)
  Neutralizing antibodies (NAb)
Explore immune response to MT-6402 treatment | 28 days (Parts 1 and 2)
  Change from baseline in immune cells
Characterize the PD profile of MT-6402 in subjects with advanced cancer | Up to 2 years (Parts 1 and 2)
  PD-L1 expression by immunohistochemistry (IHC) staining in biopsied tumor tissue, correlated with tumor response
Characterize the PD effect of MT-6402 on CMV antigen presentation | Up to 2 years (Parts 1 and 2)
  Change of CMV activated T-cells in peripheral blood
Characterize the PD effect of MT-6402 on CMV antigen presentation pre/post-dose | Up to 2 years (Part 2)
  Change in CMV activated T-cells in peripheral blood
Characterize the PD effect of MT-6402 on CMV antigen presentation | Last 2 weeks of Cycle 2 up to 2 years (Part 2)
  Comparison of tumor microenvironment
Characterize the PD effect of MT-6402 on CMV antigen presentation | Up to 2 years (Parts 1 and 2)
  Correlation between changes in CMV T-cells in peripheral blood and/or tumor biopsy with clinical response
Evaluate exposure-response relationship for MT-6402 | Up to 2 years (Parts 1 and 2)
  Change in Cmax (maximum concentration) related to clinical response
Explore relationship of circulating biomarkers with tumor response | Up to 2 years (Parts 1 and 2)
  Change in sPD-L1 levels related to PK or clinical response
Explore relationship of circulating biomarkers with tumor response | Up to 2 years (Parts 1 and 2)
  Changes in serum cytokine levels related to PK or clinical response

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - City of Hope Medical Center, Duarte, California
  - USC Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Comprehensive Care and Research Center - Atlanta, Newnan, Georgia
  - Comprehensive Care and Research Center - Chicago, Chicago, Illinois
  - University of Louisville Health - Brown Cancer Center, Louisville, Kentucky
  - Washington University School of Medicine - St. Louis, St Louis, Missouri
  - Dartmouth Hitchcock, Lebanon, New Hampshire
  - Carolina BioOncology, Huntersville, North Carolina
  - Pennsylvania Cancer Specialists and Research Institute, Gettysburg, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Sanford Cancer Center, Sioux Falls, South Dakota
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - Oncology Consultants, Houston, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas